CLINICAL TRIAL: NCT03288506
Title: Developing E-health Services (DES): The Feasibility and Acceptability of Group Based Video-conferencing for Adults With Depression
Brief Title: Developing E-health Services (DES): The Feasibility and Acceptability of Video-conferencing for Adults With Depression
Acronym: DES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Aware, Northern Ireland (Other); Northern Ireland Public Health Research Network (Other)
Responsible Party: Principal Investigator, Dr Paul Best, Lecturer, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R4773SES(DES)
Record Dates: First submitted 2017-08-16; First posted 2017-09-20 (Actual); Results first posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Population Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Google Hangout (VC) group (Experimental): This group receive peer led support for depression via Google Hangouts for 8-weeks
  Interventions: Behavioral: Google Hangout (VC) group
- Waiting list control group (No Intervention): Waiting list

INTERVENTIONS:
Behavioral: Google Hangout (VC) group — Feasibility and acceptability of online peer support groups for adults with depression. Groups will be delivered using video-conferencing technology (Google Hangouts).
  Arms: Google Hangout (VC) group

SUMMARY:
Depression impacts 1 in 5 people in the United Kingdom and is a significant risk factor for self-harming behaviours and suicide. Research has shown that those experiencing depression may feel embarrassed about seeking help from a health professional and ultimately decide not to seek support at all. This project seeks to give those people an alternative option to face-to-face support by developing a new online service using video conferencing technology. In previous studies, this technology has shown to be beneficial in treating a number of mental health problems. It may also be less expensive to run. However, as no widely available services of this type exist in the UK the full extent of potential benefits is unknown. The project seeks to answer the following questions:

* What is the likely interest in video conferencing services for depression?
* Which groups of people are likely to use the service?
* How much will this service cost?
* How much change is likely to occur when receiving therapy via video conferencing?

In order to answer these questions, Queens University Belfast are collaborating with AWARE NI, the national depression charity for Northern Ireland. Recruitment of participants who are interested in the service and delivery of the video conferencing support groups will be through AWARE NI. Results will be compared from groups that receive the video-conferencing service and those who are on a waiting list. Participants in both groups will be asked to complete surveys and take part in interviews before and after the therapy takes place. The study will have two main phases:

Phase 1: The development and in-house testing of an intervention protocol tailored towards Video Conferencing (VC) based delivery of current face-to-face peer support services. This will include interviews with facilitators, staff and current AWARE NI service users and observations of face to face groups.

Phase 2: Delivery of an 8-week group based VC support service for adults with depression. A between groups design comparing the intervention group and a waiting list control group will be used. Outcome measures will be recorded at baseline, week eight and six months using validated measures. Qualitative data in the form of interviews and fieldwork observations will also be gathered during this 8-week period.

Results will be used to inform development of a larger trial to test the effectiveness of group based video conferencing for adults with depression.

DETAILED DESCRIPTION:
Around a fifth (19%) of the UK adult population has experienced depression or depressive symptoms. The overall direct and indirect costs of treating mental illness, such as depression, are estimated at £105 billion per annum. As much as 80% of mental health care takes place in G.P surgeries or hospitals, putting increased strain on existing services and increasing pressure to find suitable alternatives. One UK based RCT investigating technology as a remote intervention for physical illness reported a 15% reduction in A&E visits, a 20% reduction in emergency admissions and an 8% reduction in tariff costs. Systematic reviews of Video-Conferencing (VC) have also shown reduced costs in relation to home care and access to on-call hospital specialists.

There is growing evidence to suggest that individuals will firstly go online for health information before seeking professional advice. As much as 4.5% of all internet searches are for health information accounting for approximately 1 out of every 20 search queries on Google. Those who seek health information online may also wish to access services however, the quality of interactive support online is questionable. A recent Cochrane review of interactive telemedicine has shown evidence of the effectiveness of VC based therapy for mental health issues. The current Secretary of State for Health has also supported the use of Skype technology as part of a 'radical redevelopment' of health services. This is in tandem with the launch of Northern Ireland's eHealth strategy in March 2016, adding to a number of policy documents suggesting this technology has the potential to increase access, lower costs and promote early intervention.

In spite of this evidence base, VC services for mental health are not widely available. As such, the full risks and benefits for clinical purposes are unknown. Several studies have shown the mental health benefits of VC as comparable with face-to-face therapy. However, the acceptability of this approach may depend on factors, such as age and technical competence. After reviewing the outcomes of VC based treatment for clients with bulimia, asserted "the distance and space provided by video therapy may have helped these clients to engage in treatment to a greater extent than would have been possible face-to face". VC has shown to be effective in the treatment of mental health conditions as well as increasing engagement for groups who would otherwise struggle to do so using face-to-face services. VC has the potential to increase access to services, target hard-to-reach groups and reduce G.P and hospital waiting times by providing alternative support mechanisms. Given the ubiquitous nature of online technologies, services are easily available and accessible which may enable preventative processes to occur sooner.

This study will address the feasibility and acceptability of group based video-conferencing support groups for adults with depression. Findings will inform the design and development of a randomised controlled trial.

Aims & objectives To test the acceptability and feasibility of delivering a peer led support group intervention for depression using VC technology.

1. To gather data sufficient to undertake a power calculation to determine the number of participants needed for a full scale RCT.
2. To explore the acceptability of randomisation within a future RCT design.
3. To establish suitability of recruitment methods.
4. To conduct a parallel qualitative study of the potential advantages and disadvantages of VC support for depression.
5. Test measures needed for economic appraisal.
6. To gather data in relation to likely interest in the service.
7. Gather preliminary evidence of the potential of the intervention to reduce depression.

Study design and methods Study design will be informed by the development and feasibility stages of the Medical Research Council (MRC) Framework for complex interventions using mixed methods. The project will involve two core phases. Phase one will focus on intervention development and in-house testing of the intervention protocol. This will include interviews and observations with facilitators, staff and current AWARE NI service users. Phase two will involve delivery of an eight week group based VC support service for adults with depression. Outcome measures for phase two will be recorded at baseline, week eight and at six months. Participants will include adults (18+) seeking support for depression. Facilitators will be AWARE NI staff and/or volunteers who are trained and experienced in delivering face to face group support meetings.

Phase 1: Intervention development, training and in-house testing During Phase 1, focus groups and interviews will be conducted with current service users to explore issues, such as the benefits of a VC support service, the barriers to accessing such a service and any suggestions regarding its current development. Member(s) of the research team at QUB will also observe face to face support groups.

In house testing will be conducted with AWARE NI staff to identify and address practical issues for example in using equipment (for example setting up cameras/speakers), logging in to the video conferencing site (Google Hangouts) as hosts and instructions needed to support staff. QUB researchers will observe staff and facilitators using the technology and interviews with staff and facilitators after testing.

Subsequently, a protocol will be produced for facilitators to complement the training programme. The manual is expected to include guidance around practical issues e.g. logging in as facilitators; checks that should be made at the start of each session (such as internet connection); alerting members as to when sessions will be beginning; checking sound issues; and informing the group if a member of the research team is observing the VC session. Guidance will also relate to dealing with drop outs and maintaining attendance records.

Current service users, staff and facilitators will be recruited through a convenience sampling method. Participant Information Sheets and Consent forms will be provided to group members through their group facilitators.

Phase 2: Intervention delivery and evaluation Approximately 4 - 6 VC groups (6-8 participants per group) will be delivered on a weekly basis for eight weeks. Groups will be facilitated peer facilitators from AWARE NI who are trained and experienced in delivering face to face support groups. Groups will be hosted securely through Google Hangouts. The online group will mirror the structure and format of face-to-face groups. Evaluation of groups will involve collection of outcome measures using validated instruments, interviews with group members/facilitators and observations of groups (described below).

Recruitment Advice was taken from the research team's statistician (Dr Chris Cardwell) and the Northern Ireland Clinical Trials Unit on sample sizes required for the feasibility study. As such, a total of 100 participants will be sought for this study.

Online support groups will be advertised as a new service by AWARE NI on the home page of the organisations website. Invitation to participate will be through an introductory page. The advertisement will specify that AWARE NI are expanding their services to include a new online support group service and that QUB will be working with AWARE NI to evaluate this new service. If participants are interested in the service and in taking part in the evaluation, they will be invited to click on a link that will lead to further information (the Participant Information Sheet). Consent will be obtained online in the first instance as a necessary step in registration and reaffirmed verbally during the VC sessions.

Registration will close once the target of 100 registers persons has been reached. Those who attempt to register after this will be advised that capacity has been reached and that they can add their name and contact details to a waiting list to be informed of when the service will become available again. This will include basic information only e.g. first name, email, age and gender. These individuals will also offered face to face support by AWARE NI outside of the study. The number of persons registering interest overall will be recorded as a measure of demand for the service and will inform the recruitment strategy of the larger RCT study.

The registration process will involve completion of several baseline measures including demographic information (first name, date of birth/age, gender, postcode, and information on any services currently receiving or accessed within the last year) and completion of validated measures of health status (see appendix A).

Randomisation Randomisation will take place following registration and completion of baseline measures (see section below). Each participant will be assigned a unique individual number and a simple random sampling procedure will be performed using online software available at http://www.randomization.com. This will result in approximately 40 participants being invited to join the VC intervention. The decision on this number was based on organisational capacity to deliver VC groups concurrently. The remaining registered participants will act as a waiting list control group (to be offered the intervention at the end of the study). A block randomisation procedure will be applied. This will involve randomly allocating in blocks of size 5 (3 to treatment and 2 to control).

Data collection Outcome measures will be recorded at baseline, week eight and six months. The research team will explore the appropriateness of the following validated instruments; Patient Health Questionnaire (PHQ-9), EQ-5D-5L measures of health outcomes and an adapted version of the Client Service Receipt Inventory (CSRI) for economic appraisal. Completion of questionnaires at each stage is expected to take approximately 5-10 minutes in total. These measurements have shown previous validity and reliability in similar studies. Feasibility will be assessed using depression outcomes; ability to recruit and retain; and fidelity (i.e. consistency of implementation across groups). Acceptability will be assessed by comparing attendance across groups, dropout rates and using through the qualitative methods (interviews and observations) specified to explore (1) reasons for taking part; and (2) user satisfaction.

Next steps

The study will inform the design and development of a large scale Randomised Controlled Trial to test the effectiveness of conducting a peer led support group intervention for depression in adults using VC technology including:

1. To investigate the effectiveness of VC based support in comparison to face-to-face support for reducing depression in adults
2. To conduct a multi-site economic appraisal of the costs and outcomes of VC support for depression.

Collaborators at AWARE and project advisors at Mindtech will advise the research team on potential UK partner organisations for the main NETS study. To date, Action on Depression (Scotland) and Depression Alliance (England) have expressed interest and support for the main NETS application.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, adults with depression (not required to have a formal diagnosis to participate), not currently an AWARE NI service user or accessed AWARE NI services in the past 12 months, a resident of Northern Ireland and not actively suicidal.

Exclusion Criteria:

* Actively suicidal, live outside Northern Ireland, currently accessing AWARE NI services or have accessed within the previous 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Best, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- AWARE NI, Belfast, Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armfield NR, Gray LC, Smith AC. Clinical use of Skype: a review of the evidence base. J Telemed Telecare. 2012 Apr;18(3):125-7. doi: 10.1258/jtt.2012.SFT101. Epub 2012 Feb 23. PMID 22362829
- [Background] Best, P., Foye, U., Taylor, B., Hazlett, D., & Manktelow, R. (2013). Online interactive suicide support services: Quality and accessibility. Mental Health Review Journal, 18(4), 226-239.
- [Background] Best, P., Manktelow, R., & Taylor, BJ. (2014). Social Work and Social Media: Online Help-Seeking and the Mental Well-Being of Adolescent Males. British Journal of Social Work. (advanced access) http://doi.org/10.1093/bjsw/bcu130
- [Background] Chong J, Moreno F. Feasibility and acceptability of clinic-based telepsychiatry for low-income Hispanic primary care patients. Telemed J E Health. 2012 May;18(4):297-304. doi: 10.1089/tmj.2011.0126. Epub 2012 Mar 16. PMID 22424078
- [Background] Centre for Mental Health (2010). The economic and social costs of mental health problems in 2009/10. Accessed 4th December 2015 from http://www.centreformentalhealth.org.uk/economic-and-social-costs
- [Background] De Las Cuevas C, Arredondo MT, Cabrera MF, Sulzenbacher H, Meise U. Randomized clinical trial of telepsychiatry through videoconference versus face-to-face conventional psychiatric treatment. Telemed J E Health. 2006 Jun;12(3):341-50. doi: 10.1089/tmj.2006.12.341. PMID 16796502
- [Background] Department Of Health. (2014). Five Year Forward View, Retrieved July, 8, 2015 from https://www.england.nhs.uk/wp-content/uploads/2014/10/5yfv-web.pdf
- [Background] Department of Health, Social Services and Public Safety. (2011a). Transforming your care: Review of health and social care in Northern Ireland. Retrieved July, 10, 2015 from http://www.dhsspsni.gov.uk/transforming-your-care-review-of-hsc-ni-final-report.pdf
- [Background] Flodgren G, Rachas A, Farmer AJ, Inzitari M, Shepperd S. Interactive telemedicine: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2015 Sep 7;2015(9):CD002098. doi: 10.1002/14651858.CD002098.pub2. PMID 26343551
- [Background] Hollis C, Morriss R, Martin J, Amani S, Cotton R, Denis M, Lewis S. Technological innovations in mental healthcare: harnessing the digital revolution. Br J Psychiatry. 2015 Apr;206(4):263-5. doi: 10.1192/bjp.bp.113.142612. PMID 25833865
- [Background] Morahan-Martin JM. How internet users find, evaluate, and use online health information: a cross-cultural review. Cyberpsychol Behav. 2004 Oct;7(5):497-510. doi: 10.1089/cpb.2004.7.497. PMID 15667044
- [Background] Simpson, S., Bell, L., Britton, P., Mitchell, D., Morrow, E., Johnston, L. A.,. . . Brebner, J. (2006). Does video therapy work? A single case series of bulimic disorders. European Eating Disorders Review, 14, 226-241.doi:10.1002/erv.686
- [Background] The Google Corporation. (2015). A remedy for your health-related questions: health info in the Knowledge Graph. Accessed December 14th 2015 at http://googleblog.blogspot.co.uk/2015/02/health-info-knowledge-graph.html.
- [Background] Wade VA, Karnon J, Elshaug AG, Hiller JE. A systematic review of economic analyses of telehealth services using real time video communication. BMC Health Serv Res. 2010 Aug 10;10:233. doi: 10.1186/1472-6963-10-233. PMID 20696073
- [Background] Yuen EK, Herbert JD, Forman EM, Goetter EM, Juarascio AS, Rabin S, Goodwin C, Bouchard S. Acceptance based behavior therapy for social anxiety disorder through videoconferencing. J Anxiety Disord. 2013 May;27(4):389-97. doi: 10.1016/j.janxdis.2013.03.002. Epub 2013 Apr 6. PMID 23764124
- [Derived] Best P, McConnell T, Davidson G, Badham J, Neill RD. Group based video-conferencing for adults with depression: findings from a user-led qualitative data analysis using participatory theme elicitation. Res Involv Engagem. 2019 Dec 5;5:40. doi: 10.1186/s40900-019-0173-z. eCollection 2019. PMID 31844555

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Google Hangout (VC) Group
Started | 60
Completed (Due to low numbers the control arm was dropped from the design and ethical amendment was sought from university committee) | 8
Not Completed | 52
Not completed — Withdrawal by Subject | 52

BASELINE CHARACTERISTICS:
Population: Descriptive statistics taken at baseline for PHQ-9 Retention is study declined rapidly after initial enrolment which meant that waiting list control was abandoned. As such, no-one entered control group
Groups:
- Control Group: This group would remain on waiting list to receive intervention at a late date
  Note: due to low retention the waiting group was not feasible and therefore results reported are intervention group only (e.g. the researchers offered intervention to those from both groups)
- Total: Total of all reporting groups
Arm/Group | Google Hangout (VC) Group | Control Group | Total
Number analyzed (Participants) | 60 | 0 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 60 |  | 60
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.1 (5.9) |  | 18.1 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 |  | 45
  Male | 15 |  | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 0 |  | 0
  More than one race | 0 |  | 0
  Unknown or Not Reported | 60 |  | 60
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 60 |  | 60
Patient Health Questionnaire (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe
  Internal consistency of the PHQ-9 has been shown to be high with Cronbach alphas of .86 and .89.
  PHQ-9 scores > 10 had a sensitivity of 88% and a specificity of 88% for Major Depressive Disorder
  Scores range from 0-27
  units on a scale | 18.1 (5.9) |  | 18.1 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire - PHQ-9
Description: Depression Measure
  PHQ-9 scores > 10 had a sensitivity of 88% and a specificity of 88% for Major Depressive Disorder.
  Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe (range of 0-27)
  Internal consistency of the PHQ-9 has been shown to be high with Cronbach alphas of .86 and .89.
Time Frame: Six months (not collected)
Population: Outcome Measure data not collected due to low study retention immediate postvention (8-weeks) and 6 months
Arm/Group | Google Hangout (VC) Group | Waiting List Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 10 months - September 2017 - June 2018
Groups:
- Waiting List Control Group: Waiting list
  Note that waiting list control group did was not implemented due to insufficient numbers
Arm/Group | Google Hangout (VC) Group | Waiting List Control Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/0
Other Adverse Events (participants affected / at risk) | 0/60 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT03288506/Prot_SAP_ICF_000.pdf